CLINICAL TRIAL: NCT02877459
Title: A Multicenter, Prospective, Single-Arm Clinical Investigation of a Modified Staged Treatment Algorithm Using the AeriSeal System - the AeriSeal-STAGE Trial
Brief Title: Clinical Investigation of a Modified Staged Treatment Algorithm Using the AeriSeal System
Acronym: STAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 630-0019
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AeriSeal System (Experimental): Subjects will be treated with AeriSeal Foam.
  Interventions: Device: AeriSeal System

INTERVENTIONS:
Device: AeriSeal System — Subjects will undergo two bronchoscopy procedures two months apart and will be treated with AeriSeal foam unilaterally, in two sub-segments during each bronchoscopy (4 segments treated in total).

SUMMARY:
A multicenter, prospective, single-arm clinical investigation to evaluate the short term and long term safety of a modified staged treatment algorithm using the AeriSeal System.

DETAILED DESCRIPTION:
The AeriSeal-STAGE trial will be a prospective, multicenter study that intends to evaluate the safety of a modified staged treatment algorithm with an escalation of dose using the AeriSeal System in the treatment of subjects with severe emphysema in a controlled trial design setting as compared to published data from prior studies. The trial is anticipated to enroll fifteen (15) study subjects with homogeneous, or upper lobe predominant heterogeneous emphysema, in three (3) centers in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide informed consent and to participate in the study
2. Subject is ≥ 40 years of age
3. Subject has a diagnosis of homogenous or heterogeneous upper lobe predominant emphysema confirmed by computerized tomography (CT) scan.
4. Subject has at least two (2) non-adjacent subsegments appropriate for treatment based upon CT scan in 2 different upper lobe segments in each lung (total 4 available subsegments)
5. Subject has clinically significant dyspnea scoring >1 on the mMRC scale of 0 - 4
6. Subject has a Six-Minute Walk Test (6MWT) distance ≥ 250 meters
7. Subject has post-bronchodilator FEV1 ≤ 45% predicted
8. Subject has Total Lung Capacity >100% predicted
9. Subject has Residual Volume >175% predicted
10. Subject has stopped smoking for at least 8 weeks prior to entering the study as confirmed by carboxyhemoglobin or cotinine levels
11. Subject has received preventive vaccinations against potential respiratory infections consistent with local recommendations or policy

Exclusion Criteria:

1. Subject has severe bullous emphysema as judged by Investigator.
2. Subject has prior lung volume reduction surgery, prior lobectomy or pneumonectomy, prior lung transplantation, prior airway stent placement, prior pleurodesis, or prior endobronchial lung volume reduction therapy of any type
3. Subject has evidence of active respiratory infection
4. Subject has an ongoing chronic obstructive pulmonary disease (COPD) exacerbation or bronchospasm
5. Subject has a known allergy to the device components:

   1. Polyether block amide - PEBAX®
   2. Polyvinyl Alcohol
   3. Glutaraldehyde
6. Subject requires ventilatory support (invasive or non-invasive)
7. Subject has diffusing capacity of the lungs for carbon monoxide (DLco) < 20% predicted
8. Subject has a post-bronchodilator FEV1 < 20% predicted
9. Subject cannot tolerate corticosteroids or relevant antibiotics
10. Subject has relevant comorbidities as judged by the Investigator, or is deconditioned and cannot tolerate the stress of post-treatment inflammatory response
11. Subject has a history of recurrent clinically significant respiratory infections, defined as three (3) or more COPD exacerbations requiring hospitalization during the year prior to enrollment
12. Subject has severe gas exchange abnormalities as defined by any one of the following:

    1. Partial pressure of arterial carbon dioxide (PaCO2) >55 mm Hg
    2. Partial pressure arterial oxygen (PaO2) <45 mm Hg on room air
    3. Peripheral capillary oxygen saturation (SpO2) < 90% on ≥ 4 L/min supplemental O2, at rest
13. Subject has Pulmonary hypertension, defined as peak systolic pressure > 45 mm Hg on echocardiogram or right heart catheterization
14. Subject use of systemic steroids >20 mg/day or equivalent and/or immunosuppressive agents in the 4 weeks prior to procedure
15. Subject unable to temporarily interrupt use of heparins or oral anticoagulants (e.g., warfarin, dicumarol) per Institutional recommendations. Note: antiplatelet drugs including aspirin and clopidogrel are permitted
16. Subject has alpha1 -antitrypsin serum level of <80 mg/kg (i.e. < 11 µmol/L) at Screening
17. Subject's CT scan indicates the presence of any the following radiologic abnormalities:

    1. Pulmonary nodule on CT scan greater than 0.8 cm in diameter [Does not apply if present for 2 years or more without increase in size or if proven benign by biopsy/positron emission tomography (PET)]
    2. Radiologic picture consistent with active pulmonary infection, e.g., unexplained parenchymal infiltrate
    3. Significant interstitial lung disease
    4. Significant pleural disease
18. Subject's baseline electrocardiogram (EKG) indicates arrhythmias or conduction abnormalities
19. Subject has high cardiac risk after undergoing cardiac risk assessment in accordance with published guidelines or ischemic heart disease, congestive heart failure, renal failure or cerebrovascular disease
20. Clinically significant asthma (reversible airway obstruction), chronic bronchitis, or bronchiectasis
21. Allergy or sensitivity to medications required to safely perform bronchoscopy and the AeriSeal System treatment under general anesthesia or conscious sedation
22. Participation in an investigational study of a drug, biologic, or device within 30 days prior to entering the study or planned during the course of the study.
23. Body mass index (BMI) < 15 kg/m2 or > 35 kg/m2
24. Female subject pregnant or breast-feeding
25. Abnormal screening laboratory test results as compared to reference lab normals at individual sites as follows:

    1. Blood urea nitrogen > 1.5 x upper limit of normal
    2. Creatinine > 1.5 x upper limit of normal
    3. Aspartate aminotransferase > 1.5 x upper limit of normal
    4. Alanine aminotransferase > 1.5 x upper limit of normal
    5. Alkaline phosphatase > 1.5 x upper limit of normal
    6. White blood cells (total) absolute < 3 x 109/L or > 1.25 x upper limit of normal
    7. Hematocrit < 34 or > 1.25 x upper limit of normal
    8. Platelets < 100 or > 450 K/µL
    9. Prothrombin time or International Normalized Ratio (INR) > 1.5 x upper limit of normal
    10. Partial thromboplastin time > 1.5x upper limit of normal
    11. Positive Beta human chorionic gonadotropin (β-HCG) Pregnancy test (if female)
26. Subject has evidence of severe disease which in the judgment of the investigator may compromise survival for the duration of the study (24 months) e.g.:

    1. Human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS)
    2. Active malignancy
    3. Stroke or Transient ischemic attack (TIA) within 12 months of Screening visit
    4. Myocardial infarction within 6 months of Screening visit
    5. Congestive heart failure within 6 months of Screening visit defined as clinical evidence of right or left heart failure or left ventricular ejection fraction < 45% on echocardiogram
27. Subject has been diagnosed with diabetes mellitus
28. Any condition that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the subject i.e., alcoholism, high risk for drug abuse or noncompliance in returning for follow-up visits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events | 3-months post treatment period
  Assessment of Serious Adverse Events (SAEs)
  To evaluate the safety of using a modified staged treatment algorithm at 3- months following the second placement of AeriSeal foam treatment in subjects with severe emphysema. The primary endpoint will be safety of AeriSeal System treatment. Safety will be assessed by monitoring the incidence of Serious Adverse Events (SAEs), during the 3-months post treatment period. Exclusively, the incidence of a prospectively specified subset of important respiratory related SAEs (COPD exacerbations requiring hospitalization or extended hospitalization, pneumonia, acute inflammatory response occurring after 30-days posttreatment, pneumothoraces), deaths and respiratory failures will be lower as compared to published data from prior studies.

SECONDARY OUTCOMES:
Forced Expiratory Volume in one second (FEV1) | Baseline, 3-months, 6-months and 12-months
  Percent mean change relative to baseline at 3-months, 6-months and 12-months for FEV1
Residual volume (RV) | Baseline, 3-months, 6-months and 12-months
  Percent mean change relative to baseline at 3-months, 6-months and 12-months for RV
Exercise capacity as assessed by six-minute walk test (6MWT) | Baseline, 3-months, 6-months and 12-months
  Absolute change relative to baseline at 3-months, 6-months and 12-months for 6MWT
Quality of life as assessed by the St George's Respiratory Questionnaire (SGRQ) | Baseline, 3-months, 6-months and 12-months
  Absolute change relative to baseline at 3-months, 6-months and 12-months for SGRQ.
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts:
  Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease)
  A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations.
Dyspnea as assessed by the Modified Medical Research Council Dyspnea Score (mMRC) | Baseline, 3-months, 6-months and 12-months
  Absolute change relative to baseline at 3-months, 6-months and 12-months for mMRC.
  The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations.
Lobar volume reduction | 3-months
  Lobar volume reduction of the treated lobes as quantified by computerized tomography (CT) scans at 3-months
Radiological signs of complications on computerized tomography (CT) scans | 3-months following the second placement of AeriSeal foam.
  Radiological signs on CT scans of complications including but not limited to pneumonias, pleural effusions and consolidation at, and outside the treatment sites and formation of lung abscesses at 3-months following the second placement of AeriSeal foam.

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Shargill, PhD, Study Director — Pulmonx Corporation
Locations (4):
- Ludwig-Boltzmann-Institut für COPD und Pneumologische Epidemiologie, Vienna, Austria
- Germany (2):
  - Charité Campus Virchow Klinikum (CVK), Berlin
  - Thoraxklinik am Universitäts klinikum Heidelberg, Heidelberg
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No